CLINICAL TRIAL: NCT03272685
Title: Impact of Very Low Nicotine Content Cigarettes in a Complex Marketplace Part of "Evaluating New Nicotine Standards for Cigarettes"
Brief Title: Impact of Very Low Nicotine Content Cigarettes in a Complex Marketplace
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Duke University (Other); University of California, San Francisco (Other); Wake Forest University (Other); University of Pennsylvania (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017NTLS107
Record Dates: First submitted 2017-08-10; First posted 2017-09-05 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Tobacco Smoking; Nicotine Dependence
Keywords: Reduced nicotine cigarettes; Alternative nicotine products; Biomarkers of tobacco exposure
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Phase III randomized, open label, multi-center study that will examine the impact of very low nicotine content (VLNC) cigarettes using an experimental marketplace that contains tobacco and nicotine products, simulating a real world environment. There are three phases: Phase 1 is smoking usual brand cigarettes. Phase 2 is access to a marketplace with usual brand cigarettes and other non-combusted nicotine and tobacco products. Phase 3 involves access to a marketplace with study cigarettes and other non-combusted nicotine and tobacco products.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Very Low Nicotine Content Cigarettes (Experimental): Very Low Nicotine Content Cigarettes (0.4 mg nicotine/g tobacco; 9 mg of tar): Median nicotine content, averaged across menthol and non-menthol cigarettes:
  Interventions: Drug: Very Low Nicotine Content Cigarettes
- Normal Nicotine Content Cigarettes (Active Comparator): Normal (Conventional) Nicotine Content (15.8 mg nicotine/g tobacco; 9 mg of tar): Median nicotine content, averaged across menthol and non-menthol cigarettes
  Interventions: Drug: Normal Nicotine Content Cigarettes

INTERVENTIONS:
Drug: Very Low Nicotine Content Cigarettes — 0.4 mg nicotine/g tobacco; 9 mg tar
  Other Names: Reduced Nicotine Content Cigarettes
  Arms: Very Low Nicotine Content Cigarettes
Drug: Normal Nicotine Content Cigarettes — 15.8 mg nicotine/g tobacco; 9 mg tar
  Other Names: Conventional Nicotine Content Cigarettes
  Arms: Normal Nicotine Content Cigarettes

SUMMARY:
This project will examine the impact of very low nicotine content (VLNC) cigarettes in a complex tobacco and nicotine product marketplace. We will compare the number of cigarettes smoked and cigarette-free days in an experimental marketplace that contains VLNC cigarettes versus normal nicotine content (NNC) cigarettes.

DETAILED DESCRIPTION:
This randomized, open label, controlled, multi-site study will simulate a "real world" tobacco environment by providing participants access to an experimental marketplace where they will be given vouchers for a specified number of points that can be exchanged for study cigarettes (varying in nicotine content described below) and non-combusted tobacco/nicotine products (smokeless tobacco, snus, electronic cigarette, medicinal nicotine replacement) and at the end of the study can exchange unspent points for money.

Subjects (N=200 in each group) will be randomly assigned to: 1) very low nicotine content cigarettes (VLNC; 0.4 mg nicotine/g tobacco) along with non-combusted tobacco/nicotine products or 2) normal nicotine content cigarettes (NNC; 15.8 mg nicotine/g tobacco) along with non-combusted tobacco/nicotine products.

Smokers will undergo an orientation visit for screening and then enter a three phase experimental trial:

1. Phase 1 - Baseline: Two week baseline assessment period during usual brand cigarette smoking.
2. Phase 2 - Marketplace Adaptation: Two week period where subjects have access to the marketplace that provides their preferred usual brand cigarettes and selected non-combusted tobacco products to allow the subject to adjust to the marketplace prior to randomization;
3. Phase 3 - Intervention: Randomization to a marketplace with access to either VLNC or NNC cigarettes plus non-combusted products for a 12 week period.

Biomarker samples are collected at baseline, end of Phase 2 and end of week Phase 3 (week 12).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female;
2. 18/21 (legal age to purchase tobacco at site);
3. Biochemically confirmed smoker.

Exclusion Criteria:

1. Unstable health condition;
2. Unstable medications;
3. Pregnant or nursing.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PHD, Principal Investigator — University of Minnesota
Locations (6):
- United States (6):
  - Tobacco Research Center, San Francisco, California
  - Tobacco Research Programs, Minneapolis, Minnesota
  - The Center for Addiction Science and Technology, Durham, North Carolina
  - Wake Forest Tobacco Control Center of Excellence, Winston-Salem, North Carolina
  - Center for Interdisciplinary Research on Nicotine Addiction, Philadelphia, Pennsylvania
  - Brown University Center for Alcohol and Addiction Studies School of Public Health, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Intend to share findings from this research through publications and presentations. Institutions and individuals wishing to access any resources or data must contact the Principal Investigator (Hatsukami). Data will be available in two formats. One will be a summary of the data, with graphs and tables, posted as pdf files and as raw individual-level data for analysis. Data generated by this grant will be made to outside investigators, according to NIH Guidance. When data are shared, there will be no limits placed on how the data will be used. Users will agree, however, that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. A record of transfer of data and a copy of the dataset that was distributed will be kept by University of Minnesota.
Time Frame: Data will not be available until primary and secondary papers are accepted for publication.
Access Criteria: Persons requesting data must do so in writing, identifying their affiliation and how the data will be used. Upon review, access will be determined.

REFERENCES:
- [Derived] Said RJ, Carroll DM, Luo X, Hu J, Cao Q, Tessier KM, Bittencourt L, Hatsukami DK; Center for Evaluation of Nicotine in Cigarettes (CENIC). Secondary analysis of a randomized clinical trial of very low nicotine cigarettes: Outcomes across social and demographic groups. Prev Med. 2025 Dec;201:108362. doi: 10.1016/j.ypmed.2025.108362. Epub 2025 Jul 21. PMID 40701191
- [Derived] Hatsukami DK, Jensen JA, Carroll DM, Luo X, Strayer LG, Cao Q, Hecht SS, Murphy SE, Carmella SG, Denlinger-Apte RL, Colby S, Strasser AA, McClernon FJ, Tidey J, Benowitz NL, Donny EC. Reduced nicotine in cigarettes in a marketplace with alternative nicotine systems: randomized clinical trial. Lancet Reg Health Am. 2024 Jun 3;35:100796. doi: 10.1016/j.lana.2024.100796. eCollection 2024 Jul. PMID 38911348

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 799 potential participants were consented and attended the screening visit. 535 eligible participants entered Phase 1; 491 continued on to Phase 2; 438 were randomized into Phase 3. See description of Phases under Study Description.
Groups:
- Very Low Nicotine Content Cigarettes: Very Low Nicotine Content Cigarettes: 0.4 mg nicotine/g tobacco; 9 mg of tar
- Normal Nicotine Content Cigarettes: Normal (Conventional) Nicotine Content: 15.8 mg nicotine/g tobacco; 9 mg of tar
Period: Overall Study
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Started | 220 | 218
Completed | 166 | 173
Not Completed | 54 | 45

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are among those who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 220 | 218 | 438
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 212 | 209 | 421
  >=65 years | 8 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 102 | 225
  Male | 97 | 116 | 213
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 6 | 7 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 45 | 54 | 99
  White | 143 | 139 | 282
  More than one race | 21 | 13 | 34
  Unknown or Not Reported | 2 | 0 | 2
Cigarettes Per Day (CPD) [Mean (Standard Deviation); unit: Number of Cigarettes Per Day] — Time Frame: Number of cigarettes smoked per day reported during Phase 2. Phase 2 CPD was used as the baseline data point.
  Number of Cigarettes Per Day | 15.6 (6.9) | 15.5 (7.6) | 15.5 (7.3)

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Day (CPD)
Description: The mean cigarettes (study and non-study cigarettes) smoked per day based on 7 days Daily Interactive Voice Response (IVR) data at the end of Phase 3 (experimental marketplace with study cigarettes) compared to Phase 2 (experimental marketplace with usual brand cigarettes).
Time Frame: 7 days prior to week 12 visit
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 168 | 173
cigarettes per day | 7.05 (7.88) | 12.95 (9.07)

2. Primary Outcome: Number of Smoke-free Days
Description: Rate of smoke-free days, defined as no cigarettes smoked in the past 24 hours calculated as the proportion of smoke-free days out of the total number of days in Phase 3.
  Number of smoke free days based on the interactive voice response (IVR)
Time Frame: day 1 of study until day before week 12 visit
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 218 | 217
days | 18.6 (28) | 5.1 (13.8)

3. Secondary Outcome: Percent Change in 2-cyanoethyl-mercapturic Acid (CEMA)
Description: Change in CEMA (biomarker for the mercapturic acid acrylonitrile) from end of Phase 2 (experimental marketplace with usual brand cigarettes) to end of Phase 3 (experimental marketplace with study cigarettes).
Time Frame: The last visit in Phase 2 is the end of the baseline
Measure: Median (Inter-Quartile Range); unit: percentage of change
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 161 | 170
percentage of change | -34 [-82 to 21] | 8 [-38 to 61]

4. Secondary Outcome: Study Cigarettes Per Day
Description: The mean study cigarettes smoked per day based on 7 days Daily Interactive Voice Response (IVR) data at the end of Phase 3 (experimental marketplace with study cigarettes) compared to Phase 2 (experimental marketplace with usual brand cigarettes).
Time Frame: 12 weeks (Phase 3) on study cigarettes
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 168 | 173
cigarettes per day | 5.33 (6.86) | 12.42 (9.23)

5. Secondary Outcome: Seven Day Point-prevalence CO-verified Abstinence
Description: Total cigarettes per day equal to 0 for all 7 days before the week 12 visit and carbon monoxide (CO) ≤ 6ppm at week 12.
Time Frame: 7 days before week 12 visit
Measure: Count of Participants; unit: Participants
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
Number analyzed (Participants) | 220 | 218
Participants | 41 | 15

ADVERSE EVENTS:
Time Frame: Adverse Events reported during Phase 3 intervention regardless of relationship, up to a total of 12 weeks.
Description: Participants were queried for any medical care, health or medication changes since their last visit.
Groups:
- Normal Nicotine Content Cigarettes: Normal (Conventional) Nicotine Content (15.8 mg/g nicotine/g tobacco; 9 mg of tar
Arm/Group | Very Low Nicotine Content Cigarettes | Normal Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/218
Serious Adverse Events (participants affected / at risk) | 7/220 | 6/218
Other Adverse Events (participants affected / at risk) | 39/220 | 42/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Nicotine Content Cigarettes (N=220) | Normal Nicotine Content Cigarettes (N=218)
Hospitalization (General disorders) | 6 (6) | 6 (6)
Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Nicotine Content Cigarettes (N=220) | Normal Nicotine Content Cigarettes (N=218)
Elevated CES-D score (Psychiatric disorders) | 39 (40) | 42 (47) — Center for Epidemiologic Studies Depression Scale
Cough (Respiratory, thoracic and mediastinal disorders) | 35 (37) | 20 (21)
Nasal congestion/Rhinorrhea (General disorders) | 34 (38) | 21 (28)
Headache/Migraine (General disorders) | 34 (38) | 17 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (29) | 22 (28)
Sore/Itchy/Irritated Throat (General disorders) | 21 (23) | 13 (16)
Irritability/Frustration (General disorders) | 20 (20) | 13 (13)
Stress (Social circumstances) | 19 (19) | 14 (16)
Depressed/Sad Mood (Psychiatric disorders) | 16 (18) | 16 (17)
Fever (General disorders) | 19 (19) | 10 (10)
Anxious/Nervous (General disorders) | 14 (14) | 14 (14)
Fatigue (General disorders) | 13 (14) | 13 (14)
Increase in Phlegm (General disorders) | 12 (12) | 11 (11)
Diarrhea (General disorders) | 14 (16) | 6 (7)
Vomiting (General disorders) | 12 (13) | 7 (7)
Toothache (General disorders) | 6 (7) | 12 (13)
Productive Cough/Lung Fullness (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 11 (11)
Insomnia (General disorders) | 11 (11) | 3 (3)
Infection (Infections and infestations) | 11 (15) | 3 (3)

LIMITATIONS AND CAVEATS:
1. Simulated natural environment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03272685/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT03272685/ICF_001.pdf